CLINICAL TRIAL: NCT01204177
Title: A Phase II Trial of BAY86-9766 Plus Sorafenib as First Line Systemic Treatment for Hepatocellular Carcinoma (HCC)
Brief Title: Assessing BAY86-9766 Plus Sorafenib for the Treatment of Liver Cancer.
Acronym: BASIL
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 14899
Record Dates: First submitted 2010-09-16; First posted 2010-09-17 (Estimated); Last update posted 2013-09-06 (Estimated); Status verified 2013-09

CONDITIONS: Carcinoma, Hepatocellular
Keywords: Hepatocellular carcinoma (HCC); MEK inhibitor; Sorafenib; Disease control rate (DCR); Safety
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Sorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm 1 (Experimental)
  Interventions: Drug: BAY86-9766 MEK Inhibitor + Sorafenib

INTERVENTIONS:
Drug: BAY86-9766 MEK Inhibitor + Sorafenib — All patients who meet the entry criteria will receive BAY86-9766 50mg (2x20mg + 1x10mg capsules) twice daily in combination with sorafenib 800 mg (2x200 mg tablets bid). During the first 3 weeks they will receive a reduced dose of sorafenib: 600 mg / daily (1x200mg tablet in the morning + 2x200mg tablets in the evening) daily. This dose will be increased to the standard dose of 800 mg (400 mg bid) if no major side effects occur. Treatment until PD or until one of the withdrawal criteria for this study is met as described in the protocol (e.g. radiological progression or clinical progression)

SUMMARY:
This study investigates the safety and efficacy of the combination therapy with BAY86-9766 and sorafenib in patients with liver cancer. Safety will be determined by laboratory and other evaluations. Efficacy of the combination BAY86-9766 and sorafenib will be determined by disease control rate, overall survival, time to progression, response rate and duration of response.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female age >/= 18 years of age
* Life expectancy >/= 12 weeks
* Histologically or cytologically confirmed diagnosis of HCC, unresectable advanced or metastatic
* Liver function status of Child-Pugh class A. Child-Pugh status based on clinical findings and laboratory results during the screening period
* Eastern Cooperative Oncology Group performance status (ECOG PS) of 0 or 1
* Patients must have at least one naïve (not previously treated by locoregional therapy) uni-dimensional measurable lesion by CT or MRI according to RECIST 1.1
* Adequate bone marrow, liver and renal function

Exclusion Criteria:

* Previous or concurrent cancer other than HCC, except for cervical carcinoma in situ, basal cell carcinoma, superficial bladder tumors.
* History of cardiac disease: Congestive heart failure (CHF), unstable angina, arrhythmias, Uncontrolled hypertension
* Clinically significant GI bleeding (CTCAE grade 3 or higher) within 30 days
* Renal failure requiring hemo- or peritoneal dialysis
* Known human immunodeficiency virus (HIV) infection
* Known history or symptomatic metastatic brain or meningeal tumors
* History of organ allograft.
* History of interstitial lung disease (ILD).
* Excluded previous therapies and medications:

  * Prior use of systemic anti-cancer treatment for HCC including cytotoxic chemotherapy, targeted agents, or any experimental therapy
  * Radiotherapy within 4 weeks prior to start of study treatment
  * Any other investigational agents within 4 weeks from the first dose of study treatment
  * Major surgery within 4 weeks of start of study
  * Concomitant use of strong inhibitors and strong inducers of CYP3A4

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2010-12; Primary Completion 2011-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Disease Control Rate (DCR) | From first dose of combination treatment until last tumor evaluation

SECONDARY OUTCOMES:
Overall Survival (OS) | 1st dose of study medication to last date of follow up
Time To Progression (TTP) | 1st dose of study medication until disease progression
Response Rate (RR) | 1st dose of study medication until last tumor evaluation
Duration Of Response (DOR) | 1st dose of study medication until last tumor evaluation
Safety: physical examination, vital signs, adverse events, safety lab | At day 1, 8, 15 of cycle 1 and 2 and day 1 of each next cycle until 30 days after EOT
Patients reported hepatobiliary cancer symptoms and Health Related Quality of Life (HRQoL) | At day 1 of each cycle and within 7 day after the last treatment
Pharmacokinetic (PK) profiles of BAY86-9766 and sorafenib to evaluate drug exposure (not in all patients) | Day -3, cycle 2 (day 1)
Biomarkers | At screening, day 1 of cycle 1 - 4, EOT

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (10):
- Hong Kong (2):
  - Shatin, New Territories
  - Hong Kong
- Singapore, Singapore
- South Korea (4):
  - Junggu, Daegu Gwang''yeogsi
  - Goyang-si, Gyeonggido
  - Busan
  - Seoul
- Taiwan (3):
  - Kaohsiung City
  - Tainan
  - Taipei

REFERENCES:
- [Derived] Lim HY, Heo J, Choi HJ, Lin CY, Yoon JH, Hsu C, Rau KM, Poon RT, Yeo W, Park JW, Tay MH, Hsieh WS, Kappeler C, Rajagopalan P, Krissel H, Jeffers M, Yen CJ, Tak WY. A phase II study of the efficacy and safety of the combination therapy of the MEK inhibitor refametinib (BAY 86-9766) plus sorafenib for Asian patients with unresectable hepatocellular carcinoma. Clin Cancer Res. 2014 Dec 1;20(23):5976-85. doi: 10.1158/1078-0432.CCR-13-3445. Epub 2014 Oct 7. PMID 25294897